CLINICAL TRIAL: NCT06596876
Title: A Randomized, Controlled, Double-blind, Double-dummy, Multicenter Phase III Study to Evaluate the Efficacy and Safety of HRG2010 in Parkinson's Disease With Motor Fluctuations
Brief Title: A Study to Evaluate the Efficacy and Safety of HRG2010 in Parkinson's Disease With Motor Fluctuations
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRG2010-301
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRG2010 and Sustained-release Carbidopa/Levodopa administered placebo (Experimental)
  Interventions: Drug: HRG2010; Sustained-release Carbidopa/Levodopa administered placebo
- Sustained-release Carbidopa/Levodopa and HRG2010 placebo (Active Comparator)
  Interventions: Drug: Sustained-release Carbidopa/Levodopa; HRG2010 placebo

INTERVENTIONS:
Drug: HRG2010; Sustained-release Carbidopa/Levodopa administered placebo — Subjects will receive HRG2010 and Sustained-release Carbidopa/Levodopa administered placebo administered orally.
  Arms: HRG2010 and Sustained-release Carbidopa/Levodopa administered placebo
Drug: Sustained-release Carbidopa/Levodopa; HRG2010 placebo — Subjects will receive Sustained-release Carbidopa/Levodopa and HRG2010 placebo administered orally.
  Arms: Sustained-release Carbidopa/Levodopa and HRG2010 placebo

SUMMARY:
The study is a multicenter, randomized, double-blind, double-dummy, active-controlled, Phase III clinical study. The aim of this trial is to evaluated the efficacy and assessed the safety of HRG2010 compared with a sustained-release cabridopa-levodopa formulation in Parkinson's Disease With Motor Fluctuations.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female who are at age 40~80 years with PD, consistent with the International Parkinson and Movement Disorder Society Clinical Diagnostic Criteria and who are being treated with stable regimens of DDCI+LD but experiencing motor fluctuations.
2. Mini Mental State Examination (MMSE) ≥ 24 at Screening Visit.
3. Hoehn and Yahr Stage I-IV when "on" at Screening Visit.
4. At Screening, the participant has predictable "Off" periods.
5. Able and willing to provide a written informed consent.

Exclusion Criteria:

1. Diagnosed with atypical or secondary parkinsonism.
2. History of narrow angle glaucoma、peptic ulcer disease or upper gastrointestinal hemorrhage.
3. Had prior functional neurosurgical treatment for PD or if such procedure(s) are planned or anticipated during the study period.
4. Nonresponsive to LD therapy.
5. In the opinion of the clinical investigator, Subjects who should not participate in the study.
6. Subjects who are allergic to the investigational drug to be used in this study.
7. Pregnant or breastfeeding.
8. Participants who have previously participated in an HRG2010 study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-02-14 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in "Off" time at Week 21 | Last three days collected at the end of treatment period, at Week 21

SECONDARY OUTCOMES:
Change from baseline in "On" Time Without Troublesome Dyskinesia at Week 21 | Last three days collected at the end of treatment period, at Week 21
Change from baseline in the Movement Disorders Society Version of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) at Week 21 | Week 21
Change from baseline in the 39-item Parkinson's Disease Questionnaire (PDQ-39) at Week 21 | Week 21
Adverse events | Week 23

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided